CLINICAL TRIAL: NCT01059903
Title: Single-site, Open-label, Randomized, Cross-over Trial to Evaluate the Bioequivalence of Single Dose Rotigotine Transdermal Patch (4.5mg/10cm2) Comparing Two Different Formulations
Brief Title: Study in Healthy Volunteers to Prove That Two Different Formulations of Rotigotine Patches Deliver Equivalent Drug Amount to the Body
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: UCB Pharma (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Basic Science
Other Study IDs: SP0987
Record Dates: First submitted 2010-01-28; First posted 2010-02-01 (Estimated); Results first posted 2011-03-03 (Estimated); Last update posted 2012-05-22 (Estimated); Status verified 2012-05

CONDITIONS: Healthy Volunteers
Keywords: Rotigotine; Neupro®; Transdermal Patch
MeSH Terms: interventions — rotigotine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Rotigotine PR2.2.1 first (Experimental): Rotigotine transdermal patch 4.5 mg/10 cm^2, test drug product PR2.2.1 followed by Rotigotine transdermal patch 4.5 mg/10 cm^2, reference drug product PR2.1.1 separated by a washout phase of at least 5 days
  Interventions: Drug: Rotigotine transdermal patch
- Rotigotine PR2.1.1 first (Experimental): Rotigotine transdermal patch 4.5 mg/10 cm^2, reference drug product PR2.1.1 followed by Rotigotine transdermal patch 4.5 mg/10 cm^2, test drug product PR2.2.1 separated by a washout phase of at least 5 days
  Interventions: Drug: Rotigotine transdermal patch

INTERVENTIONS:
Drug: Rotigotine transdermal patch — Rotigotine 4.5 mg/10 cm^2 patch applied for 24 hours
  Other Names: Neupro®

SUMMARY:
The major aim of this study is to investigate and compare the drug amount delivered to the body after sequential application of two Rotigotine patches of two different formulations

ELIGIBILITY:
Inclusion Criteria:

* Healthy White, male volunteers between 18 and 55 years of age (inclusive).
* BMI between 19 and 28 kg/m^2 (inclusive)

Exclusion Criteria:

* Previous participation in a clinical study with Rotigotine
* History or current condition of epilepsy and/or seizures
* Known clinically relevant allergy or known/suspected clinically relevant drug hypersensitivity
* History of significant skin hypersensitivity to adhesives or other transdermal products or recently unresolved contact dermatitis
* History or present condition of an atopic or eczematous dermatitis, psoriasis, and/or an active skin disease
* Clinically relevant abnormality in physical examination, ECG, vital signs or safety laboratory examinations
* Positive HIV, hepatitis B or C test or positive alcohol or drug test
* Relevant hepatic or renal dysfunction
* Intake of medication that might interfere with the test drug within 2 weeks prior to dosing

Ages: 18 Years to 55 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 50 (Actual)
Dates: Start 2010-01; Primary Completion 2010-02 (Actual); Study Completion 2010-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: UCB Clinical Trial Call Center, Study Director — +1 877 822 9493 (UCB)
Locations (1):
- Mönchengladbach, North Rhine-Westphalia, Germany

REFERENCES:
- [Derived] Elshoff JP, Timmermann L, Schmid M, Arth C, Komenda M, Brunnert M, Bauer L. Comparison of the bioavailability and adhesiveness of different rotigotine transdermal patch formulations. Curr Med Res Opin. 2013 Dec;29(12):1657-62. doi: 10.1185/03007995.2013.841666. Epub 2013 Sep 23. PMID 24006953
- See also: FDA Safety Alerts and Recalls — http://www.fda.gov/Safety/MedWatch/SafetyInformation/default.htm

RESULTS

PARTICIPANT FLOW:
Recruitment Details: A total of 50 healthy, male subjects have been randomized in order to complete the trial with at least 38 subjects qualified for the Pharmacokinetic Set (PKS). Baseline characteristics refer to the PKS which is the primary analysis set.
Pre-assignment Details: Eight subjects that fulfilled predefined criteria for patch adhesiveness were excluded from the statistical analysis on the PKS. The predefined criteria were patch adhesiveness smaller than 75% at any timepoint or an adhesiveness lower than 90% for 12 hours or more.
Groups:
- Rotigotine PR2.2.1 First: Rotigotine transdermal patch 4.5 mg/10cm^2, test drug product PR2.2.1 followed by Rotigotine transdermal patch 4.5 mg/10cm^2, reference drug product PR2.1.1 separated by a washout phase of at least 5 days
- Rotigotine PR2.1.1 First: Rotigotine transdermal patch 4.5 mg/10cm^2, reference drug product PR2.1.1 followed by Rotigotine transdermal patch 4.5 mg/10cm^2, test drug product PR2.2.1 separated by a washout phase of at least 5 days
Period: Period 1: First Intervention- 24 Hours
Arm/Group | Rotigotine PR2.2.1 First | Rotigotine PR2.1.1 First
Started | 25 | 25
Completed | 24 | 24
Not Completed | 1 | 1
Not completed — Adverse Event | 1 | 1
Period: Period 2: Washout Period (>= 5 Days)
Arm/Group | Rotigotine PR2.2.1 First | Rotigotine PR2.1.1 First
Started | 24 | 24
Completed | 24 | 24
Not Completed | 0 | 0
Period: Period 3: Second Intervention- 24 Hours
Arm/Group | Rotigotine PR2.2.1 First | Rotigotine PR2.1.1 First
Started | 24 | 24
Pharmacokinetic Set (PKS) | 18 (Six subjects who fullfilled predefined criteria for patch adhesiveness were excluded from the PKS) | 22 (Two subjects who fullfilled predefined criteria for patch adhesiveness were excluded from the PKS)
Completed | 24 | 24
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Rotigotine PR2.2.1 First | Rotigotine PR2.1.1 First | Total
Number analyzed (Participants) | 18 | 22 | 40
Age Continuous [Mean (Standard Deviation); unit: years] | 37.1 (12.6) | 35.6 (9.6) | 36.3 (11.0)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0 | 0 | 0
  Male | 18 | 22 | 40
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 0
  Not Hispanic or Latino | 18 | 22 | 40
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 0 | 0
  White | 18 | 22 | 40
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Body Mass Index (BMI) [Mean (Standard Deviation); unit: kg/m^2] | 24.42 (2.71) | 24.16 (2.75) | 24.28 (2.70)
Height [Mean (Standard Deviation); unit: meter (m)] | 1.807 (0.083) | 1.807 (0.058) | 1.807 (0.069)
Weight [Mean (Standard Deviation); unit: kilogramm (kg)] | 79.94 (11.74) | 78.88 (9.14) | 79.36 (10.26)

OUTCOME MEASURES:

1. Primary Outcome: AUC(0-tz) of Unconjugated Rotigotine
Description: The AUC(0-tz) is the area under the concentration-time curve from zero up to the last analytically quantifiable concentration.
Time Frame: 0 h (predose), 1 h, 2 h, 3 h, 4 h, 6 h, 8 h, 12 h, 16 h, 24 h (before patch removal in the morning of Day 2), 25 h, 26 h, 28 h, 30 h, 32 h, 36 h, 40 h, and 48 h
Population: Pharmacokinetic Set (PKS)
Measure: Mean (Standard Deviation); unit: ng/ mL*h
Groups:
- Rotigotine PR2.2.1: Rotigotine transdermal patch 4.5 mg/10 cm^2, test drug product PR2.2.1 ; single application of 1 patch for 24 hours
- Rotigotine PR2.1.1: Rotigotine transdermal patch 4.5 mg/10 cm^2, reference drug product PR2.1.1 ; single application of 1 patch for 24 hours
Arm/Group | Rotigotine PR2.2.1 | Rotigotine PR2.1.1
Number analyzed (Participants) | 40 | 40
ng/ mL*h | 5.2704 (3.1435) | 5.4724 (2.4755)
Statistical Analysis 1: Comparison: Rotigotine PR2.2.1 vs Rotigotine PR2.1.1; Bioequivalence testing by using the 90% Confidence Interval (CI); Test type: Non-Inferiority or Equivalence — If the 90% CI for the ratio of geometric LS-Means is included within 0.8-1.25, the patches are considered bioequivalent; ANOVA; ANOVA for log-transformed values has been used as the basis for calculation of point estimates (LS-Means) and Confidence Intervals (CIs); Ratio of geometric LS-Means = 0.9028, 90% CI 2-sided [0.8411 to 0.9690] — Bioequivalence is concluded if the 90% CIs for the ratio Treatment A/ Treatment B are fully included in the acceptance range from 0.8- 1.25 for AUC(0-tz), AUC(0-inf) and Cmax

2. Primary Outcome: Cmax of Unconjugated Rotigotine
Description: The Cmax is the maximum plasma concentration.
Time Frame: as for outcome 1
Population: Pharmacokinetic Set (PKS)
Measure: Mean (Standard Deviation); unit: ng/ mL
Arm/Group | Rotigotine PR2.2.1 | Rotigotine PR2.1.1
Number analyzed (Participants) | 40 | 40
ng/ mL | 0.26156 (0.15594) | 0.25774 (0.11184)
Statistical Analysis 1: Comparison: Rotigotine PR2.2.1 vs Rotigotine PR2.1.1; Bioequivalence testing by using the 90% Confidence Interval (CI); Test type: Non-Inferiority or Equivalence — If the 90% CI for the ratio of geometric LS-Means is included within 0.8-1.25, the patches are considered bioequivalent; ANOVA; [statistical method as in outcome 1, analysis 1]; Ratio of geometric LS-Means = 0.9506, 90% CI 2-sided [0.8833 to 1.0231] — [estimate comment as in outcome 1, analysis 1]

3. Primary Outcome: AUC(0- ∞) of Unconjugated Rotigotine
Description: The AUC(0- ∞) is the area under the plasma concentration-time curve from zero up to infinity
Time Frame: as for outcome 1
Population: Pharmacokinetic Set (PKS)
Measure: Mean (Standard Deviation); unit: ng/ mL*h
Arm/Group | Rotigotine PR2.2.1 | Rotigotine PR2.1.1
Number analyzed (Participants) | 40 | 40
ng/ mL*h | 5.36933 (3.17013) | 5.56925 (2.49370)
Statistical Analysis 1: Comparison: Rotigotine PR2.2.1 vs Rotigotine PR2.1.1; Bioequivalence testing by using the 90% Confidence Interval (CI); Test type: Non-Inferiority or Equivalence — If the 90% CI for the ratio of geometric LS-Means is included within 0.8-1.25, the patches are considered bioequivalent; ANOVA; [statistical method as in outcome 1, analysis 1]; Ratio of geometric LS-Means = 0.9046, 90% CI 2-sided [0.8437 to 0.9699] — [estimate comment as in outcome 1, analysis 1]

4. Secondary Outcome: AUC(0-tz) Norm (Apparent Dose) of Unconjugated Rotigotine
Description: The AUC(0-tz) norm (apparent dose) is the area under the plasma concentration-time curve from zero up to the last analytically quantifiable concentration normalized by apparent dose (mg).
Time Frame: as for outcome 1
Population: Pharmacokinetic Set (PKS)
Measure: Mean (Standard Deviation); unit: ng/ mL*h/ mg
Arm/Group | Rotigotine PR2.2.1 | Rotigotine PR2.1.1
Number analyzed (Participants) | 40 | 40
ng/ mL*h/ mg | 2.56504 (0.88171) | 2.66067 (1.02321)

5. Secondary Outcome: AUC(0-tz) Norm (Body Weight) of Unconjugated Rotigotine
Description: The AUC(0-tz) norm (BW) is the area under the plasma concentration-time curve from zero up to the last analytically quantifiable concentration normalized by body weight (kg).
Time Frame: as for outcome 1
Population: Pharmacokinetic Set (PKS)
Measure: Mean (Standard Deviation); unit: ng*h*kg/ mL
Arm/Group | Rotigotine PR2.2.1 | Rotigotine PR2.1.1
Number analyzed (Participants) | 40 | 40
ng*h*kg/ mL | 412.942 (239.918) | 434.101 (206.274)

6. Secondary Outcome: AUC(0- ∞) Norm (Apparent Dose)
Description: The AUC(0-inf) norm (apparent dose) is the area under the plasma concentration-time curve from zero up to infinity normalized by apparent dose (mg).
Time Frame: as for outcome 1
Population: Pharmacokinetic Set (PKS)
Measure: Mean (Standard Deviation); unit: ng/ mL*h/ mg
Arm/Group | Rotigotine PR2.2.1 | Rotigotine PR2.1.1
Number analyzed (Participants) | 40 | 40
ng/ mL*h/ mg | 2.62042 (0.88891) | 2.71397 (1.03223)

7. Secondary Outcome: AUC(0- ∞) Norm (Body Weight)
Description: The AUC(0-inf) norm (BW) is the area under the plasma concentration-time curve from zero up to infinity normalized by body weight (kg).
Time Frame: as for outcome 1
Population: Pharmacokinetic Set (PKS)
Measure: Mean (Standard Deviation); unit: ng*h*kg/ mL
Arm/Group | Rotigotine PR2.2.1 | Rotigotine PR2.1.1
Number analyzed (Participants) | 40 | 40
ng*h*kg/ mL | 420.811 (242.327) | 441.761 (207.793)

8. Secondary Outcome: Cmax, Norm (Apparent Dose) of Unconjugated Rotigotine
Description: The Cmax, norm (apparent dose) is the maximum plasma concentration normalized by apparent dose (mg).
Time Frame: as for outcome 1
Population: Pharmacokinetic Set (PKS)
Measure: Mean (Standard Deviation); unit: ng/ mL/ mg
Arm/Group | Rotigotine PR2.2.1 | Rotigotine PR2.1.1
Number analyzed (Participants) | 40 | 40
ng/ mL/ mg | 0.128863 (0.045903) | 0.126144 (0.046104)

9. Secondary Outcome: Cmax, Norm (Body Weight) of Unconjugated Rotigotine
Description: The Cmax, norm (BW) is the maximum plasma concentration normalized by body weight (kg).
Time Frame: as for outcome 1
Population: Pharmacokinetic Set (PKS)
Measure: Mean (Standard Deviation); unit: ng/ mL*kg
Arm/Group | Rotigotine PR2.2.1 | Rotigotine PR2.1.1
Number analyzed (Participants) | 40 | 40
ng/ mL*kg | 20.4935 (11.9380) | 20.4489 (9.3456)

10. Secondary Outcome: Tmax of Unconjugated Rotigotine
Description: The tmax is the time to reach maximum plasma concentration after patch application.
Time Frame: as for outcome 1
Population: Pharmacokinetic Set (PKS)
Measure: Mean (Standard Deviation); unit: hours (h)
Arm/Group | Rotigotine PR2.2.1 | Rotigotine PR2.1.1
Number analyzed (Participants) | 40 | 40
hours (h) | 16.78 (5.23) | 15.75 (5.24)

11. Secondary Outcome: Mean Residence Time (MRT) of Unconjugated Rotigotine
Description: The MRT is the mean residence time.
Time Frame: as for outcome 1
Population: Pharmacokinetic Set (PKS)
Measure: Mean (Standard Deviation); unit: hours (h)
Arm/Group | Rotigotine PR2.2.1 | Rotigotine PR2.1.1
Number analyzed (Participants) | 40 | 40
hours (h) | 18.473 (1.936) | 18.186 (2.056)

12. Secondary Outcome: Rate Constant of Elimination (λz) of Unconjugated Rotigotine
Description: The λz of unconjugated rotigotine is the rate constant of elimination.
Time Frame: as for outcome 1
Population: Pharmacokinetic Set (PKS)
Measure: Mean (Standard Deviation); unit: 1/ h
Arm/Group | Rotigotine PR2.2.1 | Rotigotine PR2.1.1
Number analyzed (Participants) | 40 | 40
1/ h | 0.162587 (0.033663) | 0.165400 (0.033405)

13. Secondary Outcome: Terminal Half-Life (t1/2) of Unconjugated Rotigotine
Description: the t1/2 of unconjugated rotigotine is the terminal half-life, calculated as t1/2=ln2/ λz.
Time Frame: as for outcome 1
Population: Pharmacokinetic Set (PKS)
Measure: Mean (Standard Deviation); unit: hours (h)
Arm/Group | Rotigotine PR2.2.1 | Rotigotine PR2.1.1
Number analyzed (Participants) | 40 | 40
hours (h) | 4.4523 (0.9701) | 4.3752 (0.9677)

14. Secondary Outcome: Apparent Total Body Clearance (CL/f) of Unconjugated Rotigotine
Description: The CL/f of unconjugated rotigotine is the apparent total body clearance.
Time Frame: as for outcome 1
Population: Pharmacokinetic Set (PKS)
Measure: Mean (Standard Deviation); unit: L/ h
Arm/Group | Rotigotine PR2.2.1 | Rotigotine PR2.1.1
Number analyzed (Participants) | 40 | 40
L/ h | 1125.11 (621.56) | 1041.47 (640.57)

15. Secondary Outcome: Apparent Dose
Description: Apparent dose of unconjugated rotigotine in mg. The apparent dose was calculated by subtraction of the determined residual content of each rotigotine patch from the nominal content of rotigotine in the patch.
Time Frame: 24 hours
Population: Pharmacokinetic Set (PKS)
Measure: Mean (Standard Deviation); unit: mg
Arm/Group | Rotigotine PR2.2.1 | Rotigotine PR2.1.1
Number analyzed (Participants) | 40 | 40
mg | 1.970 (0.637) | 2.036 (0.597)

ADVERSE EVENTS:
Time Frame: Adverse Events were collected up to 14 days after the last patch removal.
Description: Adverse Events (AEs) refer to the Safety Set (SS). The SS includes all randomized subjects who received at least 1 dose of study medication.
Arm/Group | Rotigotine PR2.2.1 | Rotigotine PR2.1.1
Serious Adverse Events (participants affected / at risk) | 0/49 | 0/49
Other Adverse Events (participants affected / at risk) | 23/49 | 26/49
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Rotigotine PR2.2.1 (N=49) | Rotigotine PR2.1.1 (N=49)
Nausea (Gastrointestinal disorders) | 4 (4) | 2 (2)
Vomiting (Gastrointestinal disorders) | 2 (2) | 1 (2)
Dyspepsia (Gastrointestinal disorders) | 2 (2) | 0
Constipation (Gastrointestinal disorders) | 0 | 1 (1)
Abdominal Pain (Gastrointestinal disorders) | 0 | 1 (1)
Gingival Bleeding (Gastrointestinal disorders) | 1 (1) | 0
Application Site Pruritus (General disorders) | 4 (4) | 5 (5)
Application Site Oedema (General disorders) | 0 | 1 (1)
Application Site Paraesthesia (General disorders) | 0 | 1 (1)
Fatigue (General disorders) | 6 (7) | 4 (4)
Thirst (General disorders) | 1 (1) | 0
Lipase Increased (Investigations) | 0 | 3 (3)
Blood Amylase Increased (Investigations) | 0 | 1 (1)
Blood Creatine Phosphokinase Increased (Investigations) | 2 (2) | 0
Alanine Aminotransferase Increased (Investigations) | 0 | 1 (1)
Blood Bilirubin Increased (Investigations) | 1 (1) | 0
Anorexia (Metabolism and nutrition disorders) | 1 (1) | 0
Pain in Jaw (Musculoskeletal and connective tissue disorders) | 1 (1) | 0
Back Pain (Musculoskeletal and connective tissue disorders) | 0 | 1 (1)
Proteinuria (Renal and urinary disorders) | 1 (1) | 0
Pharyngolaryngeal Pain (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 0 | 1 (1)
Flushing (Vascular disorders) | 0 | 1 (1)
Hot Flush (Vascular disorders) | 1 (1) | 0
Orthostatic Hypotension (Vascular disorders) | 0 | 1 (1)
Herpes Simplex (Infections and infestations) | 0 | 1 (1)
Rhinitis (Infections and infestations) | 0 | 1 (1)
Headache (Nervous system disorders) | 2 (2) | 5 (5)
Dizziness (Nervous system disorders) | 5 (7) | 4 (4)
Dizziness Postural (Nervous system disorders) | 0 | 1 (1)
Somnolence (Nervous system disorders) | 4 (4) | 0
Insomnia (Psychiatric disorders) | 1 (1) | 0
Hyperhidrosis (Skin and subcutaneous tissue disorders) | 4 (4) | 2 (2)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
UCB has > 60 days but <= 180 days to review results communications prior to public release and may delete information that is confidential and compromises ongoing studies or is considered proprietary. This restriction is not intended to compromise the objective scientific integrity of the manuscript, it being understood that results shall be published regardless of outcome.